CLINICAL TRIAL: NCT01642771
Title: A Prospective, Randomized, Open, Multi-center Phase III Clinical Study Comparing Efficacy and Safety of Sequential T-FEC and TX-XEC as Post-operative Adjuvant Chemotherapy Options for the Treatment of Triple-negative Breast Cancer
Brief Title: Comparative Study on Two Post-operative Adjuvant Chemotherapy Regimens for Treating Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Breast Cancer Clinical Study Group (Other)
Responsible Party: Principal Investigator, Zhimin Shao, MD, Dr., China Breast Cancer Clinical Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBC protocol 1.1
Record Dates: First submitted 2012-07-04; First posted 2012-07-17 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: Triple-negative Breast Cancer; Post-operative adjuvant Chemotherapy; Docetaxel; Capecitabine; Epirubicin; Cyclophosphamide; Fluorouracil
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-Fu/epirubicin/CTX following Docetaxel (Active Comparator): Docetaxel for the first 3 cycles of chemotherapy followed by 3 cycles of FEC (Fluorouracil, epirubicin and cyclophosphamide) chemotherapy
  Interventions: Drug: 5-Fu/epirubicin/CTX following Docetaxel
- Docetaxel/capecitabine followed by XEC (Experimental): Docetaxel/ capecitabine (TX) for the first 3 cycles of chemotherapy followed by 3 cycles of capecitabine/epirubicin/cyclophosphamide (XEC) chemotherapy
  Interventions: Drug: Docetaxel/capecitabine followed by XEC

INTERVENTIONS:
Drug: 5-Fu/epirubicin/CTX following Docetaxel — Cycle 1-3: Docetaxel i.v. 75mg/m2 (One cycle = 21 days); Cycle 4-6: Fluorouracil i.v. 500 mg/m2, Epirubicin i.v. 75 mg/m2, Cyclophosphamide i.v. 500 mg/m2 (One cycle = 21 days)
  Other Names: Fluorouracil: 5-Fu
  Arms: 5-Fu/epirubicin/CTX following Docetaxel
Drug: Docetaxel/capecitabine followed by XEC — Cycle 1-3: Docetaxel i.v. 75 mg/m2, Capecitabine, p.o., 1000 mg/m2，b.i.d (take Capecitabine for 2 weeks and withdraw for 1 week) (One cycle = 21 days); Cycle 4-6: Capecitabine, i.v. 1000 mg/m2, b.i.d (take for 2 weeks and withdraw for 1 week),Epirubicin, i.v. 75 mg/m2, Cyclophosphamide, i.v. 500 mg/m2 (One cycle = 21 days)
  Other Names: Capecitabine: Xeloda
  Arms: Docetaxel/capecitabine followed by XEC

SUMMARY:
Recent clinical studies showed that triple-negative breast cancer patients (ER-/PR-/HER2-) may benefit more from Capecitabine chemotherapy. However, the optimum post-operative adjuvant Capecitabine chemotherapy regimen has not been determined for Chinese population with triple-negative breast cancer. Thus it's necessary to conduct a multi-center Phase III clinical trial to verify efficacy and safety of Capecitabine in the treatment of triple-negative breast cancer. In this study, a prospective, randomized, open, multi-center Phase III clinical study was conducted to compare efficacy and safety of sequential Docetaxel followed by Fluorouracil/Epirubicin/Cyclophosphamide (FEC) and sequential Docetaxel and Capecitabine followed by Capecitabine/Epirubicin/Cyclophosphamide (XEC) as post-operative adjuvant chemotherapy in the treatment of triple-negative breast cancer in Chinese population.

DETAILED DESCRIPTION:
Post-operative adjuvant chemotherapy has been shown to improve overall survival, delay local relapse and reduce distant metastasis by multiple large-scale prospective clinical trial. In registry clinical trial for Capecitabine conducted by O Shaughnessy, it revealed that a combined chemotherapy of Capecitabine and Docetaxel achieved better outcomes compared with Docetaxel alone. And the significant effect of Capecitabine was also evidenced by CHAT trial in which Trastuzumab/Docetaxel/Capecitabine regimen was proved to perform greater than Trastuzumab/Docetaxel regimen. In addition to better outcomes, Capecitabine also showed good tolerance and safety profile. In 2009, Finnish Breast Cancer Group published their study results from FinXX clinical trial on Lancet Oncology, and in this trial, they compared the efficacy between sequential Docetaxel (3 cycles) followed by 3 cycles of Fluorouracil/Epirubicin/Cyclophosphamide (FEC) and sequential Docetaxel and Capecitabine (3 cycles) followed by 3 cycles of Capecitabine/Epirubicin/Cyclophosphamide (XEC) in lymph positive or high-risk lymph negative early-stage breast cancer patients. And their results showed a better outcome in TX-XEC regimen. 5-year follow-up analysis of this trial revealed that combined Capecitabine regimen can bring more significant clinical benefits to triple-negative breast cancer patients. Another clinical trial NO1062 released their preliminary results on comparison of AC-T and AC-XT regimens and it showed that combined Capecitabine regimen can significantly improve overall survival and this effect is more obvious in triple--negative breast cancer patients.

Based on the results of FinXX and NO1062, it's of great value to optimize combined Capecitabine regimen and clarify involved questions, such as whether the efficacy of Capecitabine is related to its treatment course or not, whether Capecitabine should be combined into current standardized chemotherapy or a sequential therapy. Also, there are still no clear conclusions on the best post-operative adjuvant chemotherapy for triple--negative breast cancer patients. Especially in Chinese population, the efficacy and safety of Capecitabine in adjuvant chemotherapy has not been well established. So it's necessary to explore reasonable dosage, safety profile and efficacy of combined Capecitabine therapy. Based on this purpose, this study is hoped to compare efficacy and safety of sequential Docetaxel followed by Fluorouracil/Epirubicin/Cyclophosphamide (FEC) and sequential Docetaxel and Capecitabine followed by Capecitabine/Epirubicin/Cyclophosphamide (XEC) as post-operative adjuvant chemotherapy in the treatment of triple-negative breast cancer in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 - 70 years old;
* Histological confirmed with unilateral invasive carcinoma (all pathological types are applicable);
* Newly diagnosed conditions allowing direct surgery without any absolute contraindication for surgery;
* No mass or microscopic tumor residue after surgery resection;
* Initiate adjuvant chemotherapy within 30 days after surgery;
* Axillary lymph node positive (including the sentinel lymph node positive and lymph node positive after axillary dissection), for example, axillary lymph node negative requires that primary tumor size must be greater than 1cm;
* Definite reports on ER/PR/Her2 receptor showing all ER/PR/Her2 negative (specific definitions: immunohistochemical detection of ER <10% tumor cells is defined as ER negative, PR <10% positive tumor cells is defined as PR-negative, Her2 is 0~1+ or 2+ but determined negative via FISH or CISH detected (no amplification) is defined as Her2 negative);
* No relevant clinical or imaging evidence of metastasis showing in the preoperative examination (M0);
* Without peripheral neuropathy;
* ECOG performance score is 0 or 1;
* Postoperative recovery was good and an interval of at least one week since the surgery is necessary;
* White blood cell count> 4 × 10^9/l, neutrophil count> 2 × 10^9/l, platelet count> 100 × 10^9/l and hemoglobin 9g/dl);
* ASAT and ALAT <1.5 folds of the upper limit of normal values, alkaline phosphatase <2.5 folds of the upper limit of normal values, total bilirubin <1.5 folds of the upper limit of normal values;
* Serum creatinine <1.5 folds of the upper limit of normal value;
* Women at childbearing age should take contraception measures during treatment;
* Cardiac function: echocardiographic examination showed LEVF> 50%;
* Informed consent form signed. -

Exclusion Criteria:

* Bilateral breast cancer or carcinoma in situ (DCIS / LCIS);
* Metastasis at any location;
* Any tumor > T4a (UICC1987) (accompanied by skin involvement, lump adhesion and fixation, inflammatory breast cancer);
* Any of ER, PR or Her-2 is positive;
* Contralateral breast clinically or radiologically suspected to be malignant but not confirmed which needs a biopsy;
* Previous neoadjuvant therapy, including chemotherapy, radiotherapy and hormone therapy;
* Previously suffering from malignant tumors (except for basal cell carcinoma and cervical carcinoma in situ), including contralateral breast cancer;
* Already enrolled into other clinical trials;
* Severe systemic disease and/or uncontrollable infection, unable to be enrolled in this study
* LEVF <50% (echocardiography);
* Suffering from severe cardiovascular and cerebrovascular diseases within six months before the randomization (such as: unstable angina, chronic heart failure, uncontrollable high blood pressure > 150/90mmHg, myocardial infarction or brain vascular accident);
* Known allergic to taxane and anthracycline agents;
* Women at childbearing age refuse to take contraception measures during the treatment and 8 weeks after completion of treatment;
* Pregnant and breast-feeding women;
* Pregnancy test showed positive results before drug administration after enrolling in to the study;
* With mental illness and cognitive impairment, unable to understand trial protocol and side effects and complete trial protocol and follow-ups (systematic evaluation is required before recruiting into this study);
* Without personal freedom and independent civil capacity.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2012-06; Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
5-year disease free survival | 5 year after the completion of chemotherapy
  Including local relapse, distant metastasis, contralateral breast cancer, second primary cancer or death from any cause

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | Within 5 years after the completion of chemotherapy
  Safety will be evaluated based on adverse events observed and the number of participants with adverse events. Blood biological tests shall also be conducted for further examination.
FACT-B scale scores as a Measure of living quality | Baseline, Week 0
  FACT-B scale scores of participants would be assessed to reflect their living quality.
5-year relapse free survival, distant disease free survival and overall survival as measures of efficacy | Within 5 years after the completion of chemotherapy
  Disease relapse shall be considered as the endpoint of relapse free survival and the period between surgery and disease relapse shall be recorded as a measure of efficacy.
  Also disease distant metastasis shall be considered as the endpoint of distant disease free survival and the period between surgery and Disease distant metastasis shall be recorded as a measure of efficacy.
FACT-B scale scores as a Measure of living quality | Week 9
  FACT-B scale scores of participants would be assessed to reflect their living quality.
FACT-B scale scores as a Measure of living quality | Week 18
  FACT-B scale scores of participants would be assessed to reflect their living quality.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, M.D., Principal Investigator — China Breast Cancer Clinical Study Group
Locations (37):
- China (37):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Pekingn Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - PLA 307 Hospital, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - The First Affi liated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - South West Hospital, Chongqing, Chongqing Municipality
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Second Affiliated Hospital of Zhongshan University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou Medical College, Shantou, Guangdong
  - Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - The Fourth Clinical Medical College of Hebei Medical University, Shijiazhuang, Hebei
  - The second affiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - The third affiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan cancer hospital affiliated to Zhengzhou university, Zhengzhou, Henan
  - Hubei General Hospital, Wuhan, Hubei
  - Xiangya Hospital Central-south University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Suzhou, Jiangsu
  - Jiangsu Province Hospital, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Third Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jinlin Cancer Hospital & Institute, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Second Affiliated Hospital of Medical College of Xi'An Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Cancer Hospital, Ürümqi, Xinjiang
  - Zhejiang First Hospital, Hangzhou, Zhejiang
  - Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

REFERENCES:
- [Background] Bria E, Nistico C, Cuppone F, Carlini P, Ciccarese M, Milella M, Natoli G, Terzoli E, Cognetti F, Giannarelli D. Benefit of taxanes as adjuvant chemotherapy for early breast cancer: pooled analysis of 15,500 patients. Cancer. 2006 Jun 1;106(11):2337-44. doi: 10.1002/cncr.21886. PMID 16649217
- [Background] Mamounas EP, Bryant J, Lembersky B, Fehrenbacher L, Sedlacek SM, Fisher B, Wickerham DL, Yothers G, Soran A, Wolmark N. Paclitaxel after doxorubicin plus cyclophosphamide as adjuvant chemotherapy for node-positive breast cancer: results from NSABP B-28. J Clin Oncol. 2005 Jun 1;23(16):3686-96. doi: 10.1200/JCO.2005.10.517. Epub 2005 May 16. PMID 15897552
- [Background] Roche H, Fumoleau P, Spielmann M, Canon JL, Delozier T, Serin D, Symann M, Kerbrat P, Soulie P, Eichler F, Viens P, Monnier A, Vindevoghel A, Campone M, Goudier MJ, Bonneterre J, Ferrero JM, Martin AL, Geneve J, Asselain B. Sequential adjuvant epirubicin-based and docetaxel chemotherapy for node-positive breast cancer patients: the FNCLCC PACS 01 Trial. J Clin Oncol. 2006 Dec 20;24(36):5664-71. doi: 10.1200/JCO.2006.07.3916. Epub 2006 Nov 20. PMID 17116941
- [Background] Piccart-Gebhart MJ, Procter M, Leyland-Jones B, Goldhirsch A, Untch M, Smith I, Gianni L, Baselga J, Bell R, Jackisch C, Cameron D, Dowsett M, Barrios CH, Steger G, Huang CS, Andersson M, Inbar M, Lichinitser M, Lang I, Nitz U, Iwata H, Thomssen C, Lohrisch C, Suter TM, Ruschoff J, Suto T, Greatorex V, Ward C, Straehle C, McFadden E, Dolci MS, Gelber RD; Herceptin Adjuvant (HERA) Trial Study Team. Trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1659-72. doi: 10.1056/NEJMoa052306. PMID 16236737
- [Background] O'Shaughnessy J, Miles D, Vukelja S, Moiseyenko V, Ayoub JP, Cervantes G, Fumoleau P, Jones S, Lui WY, Mauriac L, Twelves C, Van Hazel G, Verma S, Leonard R. Superior survival with capecitabine plus docetaxel combination therapy in anthracycline-pretreated patients with advanced breast cancer: phase III trial results. J Clin Oncol. 2002 Jun 15;20(12):2812-23. doi: 10.1200/JCO.2002.09.002. PMID 12065558
- [Background] Wardley AM, Pivot X, Morales-Vasquez F, Zetina LM, de Fatima Dias Gaui M, Reyes DO, Jassem J, Barton C, Button P, Hersberger V, Torres AA. Randomized phase II trial of first-line trastuzumab plus docetaxel and capecitabine compared with trastuzumab plus docetaxel in HER2-positive metastatic breast cancer. J Clin Oncol. 2010 Feb 20;28(6):976-83. doi: 10.1200/JCO.2008.21.6531. Epub 2009 Dec 28. PMID 20038734
- [Background] Joensuu H, Kellokumpu-Lehtinen PL, Huovinen R, Jukkola-Vuorinen A, Tanner M, Asola R, Kokko R, Ahlgren J, Auvinen P, Hemminki A, Paija O, Helle L, Nuortio L, Villman K, Nilsson G, Lahtela SL, Lehtio K, Pajunen M, Poikonen P, Nyandoto P, Kataja V, Bono P, Leinonen M, Lindman H; FinXX Study Investigators. Adjuvant capecitabine in combination with docetaxel and cyclophosphamide plus epirubicin for breast cancer: an open-label, randomised controlled trial. Lancet Oncol. 2009 Dec;10(12):1145-51. doi: 10.1016/S1470-2045(09)70307-9. Epub 2009 Nov 10. PMID 19906561
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Li J, Yu K, Pang D, Wang C, Jiang J, Yang S, Liu Y, Fu P, Sheng Y, Zhang G, Cao Y, He Q, Cui S, Wang X, Ren G, Li X, Yu S, Liu P, Qu X, Tang J, Wang O, Fan Z, Jiang G, Zhang J, Wang J, Zhang H, Wang S, Zhang J, Jin F, Rao N, Ma B, He P, Xu B, Zhuang Z, Wang J, Sun Q, Guo X, Mo M, Shao Z; CBCSG010 Study Group. Adjuvant Capecitabine With Docetaxel and Cyclophosphamide Plus Epirubicin for Triple-Negative Breast Cancer (CBCSG010): An Open-Label, Randomized, Multicenter, Phase III Trial. J Clin Oncol. 2020 Jun 1;38(16):1774-1784. doi: 10.1200/JCO.19.02474. Epub 2020 Apr 10. PMID 32275467